CLINICAL TRIAL: NCT02165631
Title: The Diurnal and Nocturnal Effect of Simbrinza and Timolol on Intraocular Pressure and Ocular Perfusion Pressure
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 14-0362; UL1TR001082 (NIH)
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension; Pigment Dispersion Syndrome; Pseudoexfoliation Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma-Related Pigment Dispersion Syndrome; Exfoliation Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A-Simbinza: Patients in Group A will receive Simbrinza (brinzolamide) 1%/0.2%, with instruction for three times daily (every 8hours) administration of the medication in both eyes for a minimum of 4 weeks and a maximum of 8 weeks of medication therapy.
- Group B-Timolol: Patients in Group B will receive Timolol 0.5%, with instructions for twice daily administration (every 12 hours) of the medication in both eyes for a minimum of 4 weeks and a maximum of 8 weeks of medication therapy.

SUMMARY:
The purpose of this research study is to hypothesize that Simbrinza will achieve a decrease in intraocular pressure and increase in ocular perfusion pressure throughout the diurnal and nocturnal periods. The primary aim of this study will be to determine the effects of Simbrinza at multiple intervals throughout a 24-hour period. The secondary aim will be to compare these to those of timolol.

DETAILED DESCRIPTION:
Intraocular pressure (IOP) is a major risk factor for the development of glaucoma. In addition, it is the only modifiable factor in the prevention and subsequent treatment of glaucomatous optic neuropathy. Most clinicians only have access to a single IOP measurement during a patient visit that may only occur once every four months. These snapshots in time are probably not adequate for the optimal management of glaucoma. Diurnal IOP curves can provide a better estimate of each patient's individual IOP variation throughout the day. However diurnal curves do not typically cover another crucial time, the nocturnal period. Glaucomatous eyes have been shown to have different IOP curves during the nocturnal period compared to healthy controls. In addition, different classes of glaucoma drugs have variable IOP lowering effects during the nocturnal hours compared to the diurnal/wake period. For example, the betablocker timolol was shown to lower IOP during daytime hours but failed to lower IOP during the nocturnal period in the habitual position. Similarly, the alpha-agonist brimonidine failed to lower IOP overnight after significantly lowering IOP during the diurnal period. On the other hand, the prostaglandin analogues, including latanoprost and travoprost, lowered IOP throughout the diurnal and nocturnal periods although nocturnal lowering appears less than the daytime hours. Therefore it is crucial to determine an accurate IOP curve for each form of medication during both wake and sleep hours.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of open angle glaucoma or ocular hypertension including pigment dispersion glaucoma and pseudoexfoliation glaucoma.
* Age ≥ 18 years, of either gender, or any race/ethnicity

Exclusion Criteria:

* Females who are currently pregnant or planning to become pregnant during the study period
* Contraindications to beta blockers (see below)
* Patients currently taking oral beta blocker therapy
* Diagnosis of any other form of glaucoma other than open-angle
* Schaffer angle grade < 2 in either eye by gonioscopy
* Intraocular surgery within 6 months or laser within 3 months
* Inability to safely discontinue all ocular medications for 6 weeks
* Patients who smoke or have irregular daily sleep patterns
* History of allergy or intolerance to topical carbonic anhydrase inhibitors, or alpha-agonists
* Patients who have started or changed glucocorticoids therapy in the last 3 months
* Patients who are currently using medical or recreational marijuana
* Any use of a non-FDA approved medication for glaucoma in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Open angle glaucoma, Ocular hypertension,Pigment dispersion glaucoma, or Pseudoexfoliation glaucoma
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure Group A | 24 hours
  The primary outcome measure will be the change in intraocular pressure and ocular perfusion pressure after 4 weeks of Simbrinza therapy at multiple time points throughout a 24-hour period.

SECONDARY OUTCOMES:
Intraocular pressure Group B | 24 hours
  The secondary outcome measure will be the change in intraocular pressure and ocular perfusion pressure after 4 weeks of timolol therapy at multiple time points throughout a 24-hour period, and how this compares to similar effects by Simbrinza.

CONTACTS AND LOCATIONS:
Overall Officials: Malik Y Kahook, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Eye Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No